CLINICAL TRIAL: NCT06516172
Title: The Bern Rehab Registry - a Prospective Cohort Study in Patients With Chronic Non-communicable Diseases Participating in a Comprehensive Rehabilitation Programme
Brief Title: The Bern Rehab Registry
Acronym: BernRehabReg
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00480
Record Dates: First submitted 2024-05-28; First posted 2024-07-23 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Cardiovascular Diseases; Musculoskeletal Diseases; Pulmonary Disease
Keywords: Rehabilitation; Prevention; Physical Function; Mental Function; Participation; Disabilities
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Musculoskeletal Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with cancer: Age 18+ years, indication for cancer rehabilitation
  Interventions: Other: Comprehensive disease-specific rehabilitation
- Patients with cardiovascular diseases: Age 18+ years, indication for cardiovascular rehabilitation
  Interventions: Other: Comprehensive disease-specific rehabilitation
- Patients with musculoskeletal diseases: Age 18+ years, indication for musculoskeletal rehabilitation
  Interventions: Other: Comprehensive disease-specific rehabilitation
- Patients with pulmonary diseases: Age 18+ years, indication for pulmonary rehabilitation
  Interventions: Other: Comprehensive disease-specific rehabilitation

INTERVENTIONS:
Other: Comprehensive disease-specific rehabilitation — Participation in (a) inpatient rehabilitation, (b) outpatient centre-based, (c) outpatient digitally-enhanced centre- and home-based, or (d) outpatient home-based digital/tele rehabilitation.
  Duration is 3 weeks for inpatient and 12 weeks for outpatient programmes.

SUMMARY:
This study examines the health outcomes of patients with long-term illnesses such as cancer, heart, lung, or musculoskeletal diseases who participate in a rehabilitation programme. The programme may involve staying in a facility (inpatient), visiting a facility (outpatient), home-based care supported by digital health tools (telerehabilitation), or a combination of facility- and home-based options.

The key health outcomes being measured include physical fitness and strength, body composition (like body fat and muscle mass), specific risk factors related to the diseases, and patients' self-reported health and experience outcomes, such as feelings of anxiety, depression, fatigue, overall quality of life, and satisfaction with the rehabilitation programme.

These measurements provide important information about the patients' lung, heart, and muscle health, as well as their mental well-being. They also help to predict the likelihood of further health complications, the chance of needing to be hospitalized again, and overall quality of life. This information is useful for improving the quality of care, tailoring future provision of rehabilitation services and long-term care for patients with chronic conditions.

Additionally, the study will provide insights into how new technologies like telerehabilitation are implemented, including how well they are adopted, followed, and accepted by patients.

DETAILED DESCRIPTION:
Background:

The global demographic landscape is shifting towards an aging population, coupled with a rise in chronic, non-communicable diseases that contribute to disability and escalating healthcare costs. Recognizing this, the World Health Organization (WHO) has identified rehabilitation as a key strategy for health in the 21st century.

Aim:

The aim of this prospective cohort study is to assess the outcomes of disease-specific comprehensive rehabilitation programmes at a tertiary referral center to improve the quality of care and formulate novel research questions.

Methods:

Consecutive patients with cancer, cardiovascular, musculoskeletal, or pulmonary diseases, referred for comprehensive rehabilitation to the Centre for Rehabilitation & Sports Medicine (two locations - Berner Reha Centre and Inselspital) of the Insel Group, Bern, Switzerland, will be included. Patients will be counselled by trained advanced practice nurses, and type of delivery of the rehabilitation programme will be based on medical needs and patient preferences. Three-week inpatient programmes are performed at the Berner Reha Centre and Inselspital. Twelve-week outpatient programmes are performed at the Inselspital and delivered as centre-based, digitally-enhanced centre- and home-based, or home-based digital/tele rehabilitation.

Outcome assessments will be based on the framework of the International Classification of Functioning, Disability, and Health (ICF) of the World Health Organisation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older with a chronic non-communicable disease
* Signed general informed consent
* Referral to a comprehensive disease-specific rehabilitation program

Exclusion Criteria:

* Refuted or missing general informed consent for further use of health-related data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic, non-communicable diseases participating in a comprehensive disease-specific rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Short-term change (absolute and percentage) in cardiorespiratory fitness, measured as peak oxygen uptake (ml/min/kg) or 6 minute walking test (m) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes)
  Stratified by type of delivery and cohort
Long-term change (absolute and percentage) in cardiorespiratory fitness, measured as peak oxygen uptake (ml/min/kg) or 6 minute walking test (m) | From discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) to one year follow-up
  Stratified by type of delivery and cohort

SECONDARY OUTCOMES:
Short- and long-term change (absolute and percentage) in muscle strength, measured by grip strength (kg) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term change (absolute and percentage) in muscle mass index, measured by body impedance analysis (kg/height2) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term change (absolute and percentage) in the Extended Barthel Index (EBI, range from 0 to 64) or the Functional Independence Measure (FIM, range from 0 to 126), higher values indicate better levels physical and/or mental functioning | From rehabilitation entry to discharge (3 weeks) and from discharge to one year follow-up
  In patients participating in inpatient rehabilitation, stratified by cohort
Short- and long-term changes (absolute and percentage) in markers of anxiety, measured by Generalized Anxiety Disorder-7 questionnaire score (range from 0 to 21, higher values indicate more severe anxiety) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in markers of depression, measured by Patient Health Questionnaire-9 score (range from 0 to 27, higher values indicate more severe depression) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in markers of health-related quality of life, measured by Kansas City Cardiomyopathy Questionnaire-23 score (range from 0 to 100, higher values indicate better QoL) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  In patients with heart failure, stratified by type of delivery
Short- and long-term changes (absolute and percentage) in markers of health-related quality of life, measured by HearQoL questionnaire score (range from 0 to 3, higher values indicate better QoL) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  In patients with heart disease participating in outpatient cardiac rehabilitation or telerehabilitation
Short- and long-term changes (absolute and percentage) in markers of health-related quality of life, measured by MacNew questionnaire score (range 0 to 7, higher values indicate better QoL) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  In patients with heart disease participating in inpatient cardiac rehabilitation
Short- and long-term changes (absolute and percentage) in markers of health-related quality of life, measured by Chronic Respiratory Disease Questionnaire score (range 1 to 7, higher values indicate better QoL) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  In patients with pulmonary disease, stratified by type of delivery
Short- and long-term changes (absolute and percentage) in markers of health-related quality of life, measured by Functional Assessment of Cancer Therapy-General questionnaire score (range 1 to 5, higher values indicate better QoL) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  In patients with cancer, stratified by type of delivery
Short- and long-term changes (absolute and percentage) in office systolic blood pressure (mmHg) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in LDL-cholesterol (mmol/l) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in HbA1c (percentage) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Composite outcome, stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in hsCRP (mg/l) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in body mass index (kg/m2) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in body fat, assessed by body impedance analysis (%) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in steps per day, assessed by wrist-worn accelerometer (n) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in smoking status, assessed by questionnaire (current, former, non-smoker) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Composite outcome, stratified by type of delivery and cohort
Short- and long-term changes (absolute and percentage) in adherence to guideline-directed medical therapies (percentage of recommended medical substances taken) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and from discharge to one year follow-up
  Stratified by type of delivery and cohort
Return to work (yes, no) | At rehabilitation discharge (3 weeks for inpatient, 12 weeks for outpatient programmes) and at one year follow-up
  Stratified by type of delivery and cohort

OTHER OUTCOMES:
Time trends of proportion of patient participating in digitally-enhanced or digital/telerehabilitation (percentage) | 12 months
  Stratified by type cohort
Assessment of patient reported experience measures (PREMS) by a self-designed questionnaire on satisfaction with the rehabilitation programme (range 1 to 10, higher values indicate higher satisfaction) | From rehabilitation entry to discharge (3 weeks for inpatient, 12 weeks for outpatient programmes)
  Stratified by type of delivery and cohort

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Wilhelm, MD, Principal Investigator — Centre for Rehabilitation & Sports Medicine, Insel Group
Locations (2):
- Switzerland (2):
  - Berner Reha Centre, Centre for Rehabilitation & Sports Medicine, Insel Group, Heiligenschwendi, Canton of Bern
  - Reha Inselspital, Bern University Hospital, Centre for Rehabilitation & Sports Medicine, Insel Group, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the Centre for Rehabilitation & Sports Medicine, Insel Group Bern — http://www.rehasportmedizin.insel.ch